CLINICAL TRIAL: NCT01292135
Title: A Phase 1b, Multicenter, Open-label, Parallel-group Safety Study of a Bruton's Tyrosine Kinase (Btk) Inhibitor, PCI 32765, in Combination With Chemotherapy in Subjects With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Safety and Tolerability Study of PCI-32765 Combined With Fludarabine/Cyclophosphamide/Rituximab (FCR) and Bendamustine/Rituximab (BR) in Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1108-CA; PCI-32765 (Other: Pharmacyclics)
Record Dates: First submitted 2011-02-02; First posted 2011-02-09 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Lymphoma, B-Cell; Leukemia, Lymphoid; Leukemia, B-Cell; Bruton's Tyrosine Kinase
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Leukemia, Lymphoid; Leukemia, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCI-32765 plus fludarabine/cyclophosphamide/rituximab (FCR) (Experimental)
  Interventions: Drug: PCI-32765
- PCI-32765 plus bendamustine/rituximab (BR) (Experimental)
  Interventions: Drug: PCI-32765

INTERVENTIONS:
Drug: PCI-32765 — 420 mg daily

SUMMARY:
The purpose of this study is to establish the safety of orally administered PCI-32765 in combination with fludarabine/cyclophosphamide/rituximab (FCR) and bendamustine/rituximab (BR) in patients with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma(SLL).

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, parallel-group, nonrandomized, multicenter study of PCI 32765 420 mg once daily oral (PO) administration in combination with 2 different chemotherapy regimens in subjects with relapsed/refractory chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CLL or SLL and satisfying at least 1 of the following criteria for requiring treatment:

   * Progressive splenomegaly and/or lymphadenopathy identified by physical examination or radiographic studies
   * Anemia (<11 g/dL) or thrombocytopenia (<100,000/μL) due to bone marrow involvement
   * Presence of unintentional weight loss > 10% over the preceding 6 months
   * NCI CTCAE Grade 2 or 3 fatigue
   * Fevers > 100.5° or night sweats for > 2 weeks without evidence of infection
   * Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of < 6 months
2. 1 to 3 prior treatment regimens for CLL/SLL
3. ECOG performance status of ≤ 1
4. ≥ 18 years of age
5. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
6. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Exclusion Criteria:

1. Any chemotherapy, therapeutic antineoplastic antibodies (not including radio- or toxin immunoconjugates), radiation therapy, or experimental antineoplastic therapy within 4 weeks of first dose of study drug
2. Radio- or toxin-conjugated antibody therapy within 10 weeks of first dose of study drug
3. Concomitant use of medicines known to cause QT prolongation or torsades de pointes
4. Transformed lymphoma or Richter's transformation Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of PCI-32765 PO, or put the study outcomes at undue risk
5. Any of the following laboratory abnormalities: oAbsolute neutrophil count (ANC) < 1000 cells/mm3 (1.0 x 109/L) oPlatelet count < 50,000/mm3 (50 x 109/L) oSerum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) ≥ 3.0 x upper limit of normal (ULN) oCreatinine > 2.0 x ULN or creatinine clearance < 40 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Graef, MD, Study Director — Pharmacyclics LLC.
Locations (6):
- United States (6):
  - Dana Farber Cancer Center, Boston, Massachusetts
  - CLL Research and Treatment Program, New Hyde Park, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson, Houston, Texas

REFERENCES:
- [Derived] Brown JR, Barrientos JC, Barr PM, Flinn IW, Burger JA, Tran A, Clow F, James DF, Graef T, Friedberg JW, Rai K, O'Brien S. The Bruton tyrosine kinase inhibitor ibrutinib with chemoimmunotherapy in patients with chronic lymphocytic leukemia. Blood. 2015 May 7;125(19):2915-22. doi: 10.1182/blood-2014-09-585869. Epub 2015 Mar 9. PMID 25755291
- See also: www.pharmacyclics.com — http://www.pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Groups:
- PCI-32765 Plus Fludarabine/Cyclophosphamide/Rituximab (FCR): PCI-32765: 420 mg daily
  FCR:
  * Rituximab: 375 mg/m2 on Day 1 of Cycle 1 and a dose of 500 mg/m2 on Day 1(Cycle 2 to Cycle 6).
  * Fludarabine: 25 mg/m2/day for 3 days (Days 1 to 3) of each cycle
  * Cyclophosphamide: 250 mg/m2/day for 3 days (Days 1 to 3) of each cycle (Up to 6 Cycle)
- PCI-32765 Plus Bendamustine/Rituximab (BR): PCI-32765: 420 mg daily
  BR:
  * Rituximab: 375 mg/m2 on Day 1 of Cycle 1 and a dose of 500 mg/m2 on Day 1 (Cycle 2 to Cycle 6).
  * Bendamustine; 70 mg/m² on Day 1 and 2 of each cycle (Up to 6 Cycles)
Period: Overall Study
Arm/Group | PCI-32765 Plus Fludarabine/Cyclophosphamide/Rituximab (FCR) | PCI-32765 Plus Bendamustine/Rituximab (BR)
Started | 3 | 30
Completed | 3 | 21
Not Completed | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCI-32765 Plus Fludarabine/Cyclophosphamide/Rituximab (FCR) | PCI-32765 Plus Bendamustine/Rituximab (BR) | Total
Number analyzed (Participants) | 3 | 30 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (1.53) | 61.3 (9.58) | 60.8 (9.24)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 19 | 22
  >=65 years | 0 | 11 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 3 | 25 | 28
Region of Enrollment [Number; unit: participants]
  United States | 3 | 30 | 33

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Prolonged Hematologic Toxicity Started in Cycle 1
Time Frame: From First day of dose to 30 days after last dose of any study medication. Participants were followed with a median follow-up time of 15.8 months.
Population: The FCR arm was discontinued due to very limited use of this chemo regimen in this setting, statistical analysis were limited due to the small numbers of subjects in this treatment arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- PCI-32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR): PCI-32765: 420 mg daily
Arm/Group | PCI-32765 Plus Bendamustine/Rituximab (BR) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR)
Number analyzed (Participants) | 30 | 3
Percentage of Participants | 0 [0 to 11.6] | 0 [NA to NA] — Dispersion not calculated due to small sample size n=3.

2. Secondary Outcome: Incidence of Adverse Events Requiring Dose Delay or Discontinuation of Ibrutinib
Time Frame: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- PCI-32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR): PCI- 32765: 420 mg daily
Arm/Group | PCI-32765 Plus Bendamustine/Rituximab (BR) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR)
Number analyzed (Participants) | 30 | 3
Percentage of Participants | 53.3 | 33.3

3. Secondary Outcome: Overall Incidence of Grade ≥3 Adverse Events (AEs) Per NCI CTCAE V4.0
Time Frame: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | PCI-32765 Plus Bendamustine/Rituximab (BR) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR)
Number analyzed (Participants) | 30 | 3
Percentage of Participants | 66.7 | 0

4. Secondary Outcome: Overall Incidence of Serious Adverse Events (SAEs)
Time Frame: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | PCI-32765 Plus Bendamustine/Rituximab (BR) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR)
Number analyzed (Participants) | 30 | 3
Percentage of Participants | 20 | 33.3

5. Secondary Outcome: Overall Response Rate (Complete Response [CR] + Complete Response With Incomplete Marrow Recovery [CRi] + Nodular Partial Response [nPR] + Partial Response [PR])
Description: Response criteria are as outlined in the IWCLL 2008 criteria (Hallek 2008) and as assessed by investigator, e.g. response requires 50% reduction in lymph node size. Assessment of response to treatment will be done every 2 cycles for the first 6 months and then every 3 months thereafter until disease progression or prior to the administration of a new anticancer therapy and at follow-up visits.
Time Frame: From first response assessment to last response assessment. Participants were followed with a median follow-up time of 15.8 months.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PCI-32765 Plus Bendamustine/Rituximab (BR) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR)
Number analyzed (Participants) | 30 | 3
Percentage of Participants | 93.3 [77.9 to 99.2] | 100 [NA to NA] — Dispersion not calculated due to small sample size n=3.

6. Secondary Outcome: Sustained Hematologic Improvement in Subjects With Neutropenia, Anemia, or Thrombocytopenia at Baseline
Time Frame: as for outcome 5
Population: No participants in the FCR group had neutropenia, anemia or thrombocytopenia at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PCI-32765 Plus Bendamustine/Rituximab (BR) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR)
Number analyzed (Participants) | 30 | 0
Percentage of Participants | 76.2 [52.8 to 91.8] |

7. Secondary Outcome: Progression Free Survival Rate at 12 Months
Description: Criteria for progression are as outlined in the IWCLL 2008 criteria (Hallek 2008) and as assessed by investigator, e.g. progression defined as a 50% increase in lymph node size.
Time Frame: From first dose of any study medication to 12 months after first dose to progressive disease or death or the last clinical assessment before receiving new anticancer therapy or loss to follow-up, whichever occured the earliest.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- PCI- 32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR): PCI-32765: 420 mg daily
Arm/Group | PCI-32765 Plus Bendamustine/Rituximab (BR) | PCI- 32765 Plus Fludarabine/ Cyclophosphamide/ Rituximab (FCR)
Number analyzed (Participants) | 30 | 3
Percentage of Participants | 85.9 [66.7 to 94.5] | 100 [100 to 100]

ADVERSE EVENTS:
Groups:
- PCI-32765 Plus Fludarabine/ Cyclophosphamide/Rituximab (FCR): PCI-32765: 420 mg daily
Arm/Group | PCI-32765 Plus Bendamustine/Rituximab (BR) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/Rituximab (FCR)
Serious Adverse Events (participants affected / at risk) | 6/30 | 1/3
Other Adverse Events (participants affected / at risk) | 30/30 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 Plus Bendamustine/Rituximab (BR) (N=30) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/Rituximab (FCR) (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 Plus Bendamustine/Rituximab (BR) (N=30) | PCI-32765 Plus Fludarabine/ Cyclophosphamide/Rituximab (FCR) (N=3)
Neutropenia (Blood and lymphatic system disorders) | 12 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Conjuctivitis (Eye disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 1
Nausea (Gastrointestinal disorders) | 20 | 2
Constipation (Gastrointestinal disorders) | 9 | 0
Vomiting (Gastrointestinal disorders) | 9 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Tongue ulcerlation (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 14 | 0
Oedema peripheral (General disorders) | 10 | 0
Pyrexia (General disorders) | 7 | 0
Chills (General disorders) | 5 | 0
Asthenia (General disorders) | 3 | 0
Pain (General disorders) | 3 | 0
Chest discomfort (General disorders) | 2 | 0
Impaired healing (General disorders) | 2 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0
Seasonal allergy (Immune system disorders) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 1
Sinusitis (Infections and infestations) | 8 | 0
Urinary tract infection (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Pneomonia (Infections and infestations) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 6 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 0
Weight decreased (Investigations) | 3 | 0
Blood uric acid increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3
Fluid retention (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Headache (Nervous system disorders) | 9 | 0
Dizziness (Nervous system disorders) | 7 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 7 | 0
Depression (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 3 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash maculo papular (Skin and subcutaneous tissue disorders) | 5 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Sunburn (Skin and subcutaneous tissue disorders) | 2 | 0
Flushing (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Oral herpes (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1
Skin Infection (Infections and infestations) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No